CLINICAL TRIAL: NCT04588025
Title: Disposable Perfusion Phantom for Accurate DCE (Dynamic Contrast Enhanced)-MRI Measurement of Pancreatic Cancer Therapy Response
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Harrison Kim, Associate Professor, Division of Advanced Medical Imaging Research, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB- 300003007
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The healthy group is going to be the group to establish a baseline for the pancreatic group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Healthy Volunteers (Active Comparator)
  Interventions: Device: Point-of-care Portable Perfusion Phantom, P4
- Pancreatic Cancer Participants (Active Comparator)
  Interventions: Device: Point-of-care Portable Perfusion Phantom, P4

INTERVENTIONS:
Device: Point-of-care Portable Perfusion Phantom, P4 — P4 is a perfusion phantom developed by Dr. Harrison Kim that can significantly reduce variation in quantitating perfusion of human abdominal tissues across MRI scanners.

SUMMARY:
The goal of this study is to investigate whether the therapeutic response of pancreatic tumors can be accurately assessed using quantitative DCE-MRI, when the inter/intra-scanner variability is reduced using the Point-of-care Portable Perfusion Phantom, P4. The intra-scanner variability over time leads to errors in therapy monitoring, while the inter-scanner variability impedes the comparison of data among institutes. The P4 is small enough to be imaged concurrently in the bore of a standard MRI scanner with a patient for real-time quality assurance. The P4 is safe, inexpensive and easily operable, thus it has great potential for widespread and routine clinical use for accurate diagnosis, prognosis and therapy monitoring.

This study has identified two arms, one arm is healthy individuals that will undergo DCE MRI at three different MRI locations to establish baseline results. The healthy volunteers will undergo these MRIs prior to the second arm, which contains patients with pancreatic cancer. The pancreatic cancer patients will only have DCE MRI done at one location.

ELIGIBILITY:
Healthy Volunteer - a small number of healthy volunteers (5) will be used as the control group.

Inclusion Criteria:

* Targeted/planned enrollment in the study will include all racial/ethnic groups with no groups excluded on the basis of race, ethnicity or gender.
* Participants should be 19 years of age or older
* Participants should not have any known major health problems including but not limited to cancers, heart diseases, diabetes, high blood pressure and/or cholesterol, stroke, respiratory problems, and arthritis.

Exclusion Criteria:

* Participants having any known major health problems will be excluded.
* Participants with safety contraindications to MRI examination (determined by standard clinical screening).
* Participants on hemodialysis or with acute renal failure will be excluded. (Participants on hemodialysis and those with renal failure who receive intravenous gadolinium may be at increased risk for a condition called Nephrogenic systemic fibrosis/ Nephrogenic fibrosing dystrophy and thus will be excluded.)
* Participants may not be pregnant or lactating.
* Participants may not father a child while on this study as the treatment may indirectly affect an unborn child.
* Unless participants cannot have children because of surgery or other medical reasons, participants must have been using an effective form of birth control before starting the study.
* Participants must also agree to continue to use an effective form of birth control for 6 months after taking the study. Effective birth control includes birth control pills, patch, IUD (intrauterine device), condom, sponge, diaphragm with spermicide, or avoiding sexual activity that could cause pregnancy.

Pancreatic Cancer Participants:

Inclusion Criteria:

* Patients having biopsy proven locally advanced pancreatic cancer will be asked to participate in this study.
* Targeted/planned enrollment in the study will include all racial/ethnic groups, with no groups excluded on the basis of race, ethnicity or gender.
* Participants should be 19 years of age or older.

Exclusion Criteria:

* Participants with safety contraindications to MRI examination (determined by standard clinical screening).
* Participants on hemodialysis or with acute renal failure will be excluded.
* Participants on hemodialysis and those with renal failure who receive intravenous gadolinium may be at increased risk for a condition called Nephrogenic systemic fibrosis/ Nephrogenic fibrosing dystrophy and thus will be excluded.
* Participants may not be pregnant or lactating.
* Participants may not father a child while on this study as the treatment may indirectly affect an unborn child.
* Unless participants cannot have children because of surgery or other medical reasons, participants must have been using an effective form of birth control before starting the study.
* Participants must also agree to continue to use an effective form of birth control for 6 months after taking the study. Effective birth control includes birth control pills, patch, IUD, condom, sponge, diaphragm with spermicide, or avoiding sexual activity that could cause pregnancy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of quantitative DCE-MRI measurement with MRI 1. | Baseline
  This outcome is assigned to the 5 healthy volunteers that we will be evaluated on 3 different MRIs. Two scans will be done to establish baseline measures.
Reproducibility of quantitative DCE-MRI measurement with MRI 2. | Baseline to 3-days (MRI number 2)
  This outcome is assigned to the 5 healthy volunteers that we will be evaluated on 3 different MRIs.
Reproducibility of quantitative DCE-MRI measurement with MRI 3. | Baseline to 7-days (MRI number 3)
  This outcome is assigned to the 5 healthy volunteers that we will be evaluated on 3 different MRIs.
Measure change in blood flow within the pancreatic cancer as measured by the P4. | Baseline
  This is being done before therapy has been initiated and is being measured by the P4 during an MRI scan. The results will help determine if undergoing therapy is effective by measuring the change in blood flow and help to decide if we need to continue the current therapy or change to a different one. Blood flow often serves as a critical indicator showing a disease status.
Measure change in blood flow within the pancreatic cancer as measured by the P4. | 6 weeks post-therapy
  This is being done after therapy has been initiated and is being measured by the P4 during an MRI scan. The results will help determine if undergoing therapy is effective by measuring the change in blood flow and help to decide if we need to continue the current therapy or change to a different one. Blood flow often serves as a critical indicator showing a disease status.

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Kim, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
To be determined